CLINICAL TRIAL: NCT02064777
Title: Tacrolimus Disposition in Pediatric Transplantation: Influence of Age, Genetic Polymorphisms, Intestinal and Hepatic Relative Contribution on Pharmacokinetics, in Relationship With Clinical Outcomes
Brief Title: Prospective Tacrolimus Pharmacokinetics Study in Pediatric Living Donor Liver Transplantation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2012MAR19
Record Dates: First submitted 2014-02-14; First posted 2014-02-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-02

CONDITIONS: Pediatric Liver Transplantation
MeSH Terms: interventions — Tacrolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tacrolimus (Experimental)
  Interventions: Drug: Tacrolimus

INTERVENTIONS:
Drug: Tacrolimus

SUMMARY:
Our first aim is thus to investigate, retrospectively first and then prospectively, in de novo pediatric (living donor) liver recipients, the tacrolimus in vivo and in vitro metabolism and its variability with focus on pharmacokinetics, pharmacodynamics, and pharmacogenomics and its evolution according to the age and transplant delay. Our second aim is then to find better tacrolimus exposure markers for therapeutic drug monitoring (TDM) such as Area Under the time-concentration Curve (AUC) or intralymphocytic (PBMCs) tacrolimus concentration and a way to model and predict it without invasive tests in pediatric patients.

The final objective should be then to implement these findings in a more individualized and comprehensive immunosuppression protocol and monitoring in order to maintain adequate and well-balanced immunosuppression (preventing graft rejection while avoiding acute and long-term side effects). This is particularly important for a pediatric population exposed throughout their life to immunosuppressants.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0 to 18 years
* First Liver transplantation
* Children eligible to receive tacrolimus post transplantation
* Consent from parents

Exclusion Criteria:

* Multiorgan transplantation
* Retransplantation
* ABO incompatible donors (unless if recipients is<1 year and anti-AB antibodies are <1/32)
* Multi organ failure
* Need for additionnal therapy except for methylprednisolone to treat rejection
* Intravenous tacrolimus
* First tacrolimus administration postponed after day 3

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2013-07; Primary Completion 2014-06 (Estimated); Study Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Area Under the Time Concentration curve | day 2-day 4; day 10-day 1; > day 21

SECONDARY OUTCOMES:
Intralymphocytic tacrolimus concentration | Day 3

CONTACTS AND LOCATIONS:
Locations (1):
- Cliniques Universitaires St-Luc, Brussels, Belgium